CLINICAL TRIAL: NCT04998942
Title: Virtual Cardiac Wellness Program Following Hypertensive Disorders of Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Amy A. Sarma, MD, Cardiologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021P001285
Record Dates: First submitted 2021-07-12; First posted 2021-08-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hypertension in Pregnancy; Gestational Hypertension; Preeclampsia; Chronic Hypertension With Pre-Eclampsia; Eclampsia; Chronic Hypertension in Obstetric Context
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Intervention Model Description: In this study, we are testing different strategies to help women keep their heart healthy after a pregnancy complicated by hypertension.
  Participants may or may not undergo some of the following study procedures:
  * Complete surveys which could include topics related to activity, stress, nutrition, heart disease etc. with study staff via telephone or a secure online platform
  * Be contacted by study staff once monthly to collect subjects' weight, blood pressure, whether they are breastfeeding, exercise routine, smoking status, and stress levels
  * Meet with a nutritionist
  * Meet with an exercise physiologist
  * Participate in optional group sessions
  * Receive infographics which could include topics such as mindful living and lifestyle, prevention of heart disease, nutrition, heart disease, etc.
  Arm assignment and a description of the arms will be disclosed to participants after study completion.
Who Masked: Participant
Masking Description: In order to enable us to conduct a placebo-controlled study, we will not disclose to participants which intervention they have been assigned to. In order to obtain blinded data, incomplete disclosure is necessary to make the research scientifically valid and feasible. Unblinding subjects increases the risk that a favorable outcome is associated with the intervention simply because subjects are aware that they received an intervention and thus performing a placebo-controlled trial is necessary to determine the true effect of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Behavioral: virtual cardiac wellness program
- Placebo comparator (Placebo Comparator)
  Interventions: Behavioral: Placebo comparator

INTERVENTIONS:
Behavioral: virtual cardiac wellness program — Participants assigned to this arm will participate in the experimental intervention.
  Arms: Experimental
Behavioral: Placebo comparator — Participants assigned to this arm will participate in a placebo intervention.
  Arms: Placebo comparator

SUMMARY:
Hypertensive disorders of pregnancy (HDP) are now well-recognized risk factors for adverse outcomes in the postpartum period and for development of future cardiovascular disease (CVD). Postpartum BMI has emerged as a strong predictor of both short- and long-term blood pressure (BP) control in observational studies suggesting that earlier postpartum lifestyle modifications may be instrumental in future CVD risk reduction in women with HDP. While such lifestyle modifications are recognized as critical for postpartum health, implementation and engagement of postpartum women remains a challenge as new mothers face greater barriers to in-person care given childcare responsibilities. The proposed study will investigate the acceptability of a virtual cardiac wellness program and its impact on weight, lifestyle modifications, cardiometabolic health, patient engagement, and outcomes following HDP as compared to the standard of care for postpartum women at Massachusetts General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Women with a diagnosis of HDP inclusive of gestational hypertension, preeclampsia, eclampsia, and chronic hypertension with superimposed preeclampsia
* Pre-pregnancy BMI >18.5
* Age ≥ 18 years
* Access to a phone
* Delivery at MGH and receive longitudinal obstetrics care at MGH

Exclusion Criteria:

* Moderate or severe cognitive impairment
* Current incarceration
* Pre-pregnancy BMI ≤ 18.5
* Women without a documented pre-natal weight or weight recorded 1 year prior to pregnancy
* Baseline exercise of > 150 minutes/ week at the time of study enrollment
* Not cleared for exercise by primary OB

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Postpartum weight loss at 6 months postpartum | 1 year
  Postpartum weight loss (Last prenatal visit weight- weight at 6 months postpartum) as a proportion of weight gained during pregnancy (Last prenatal visit weight- either 1st prenatal weight or pre-pregnancy weight within 1 year)

SECONDARY OUTCOMES:
Postpartum weight loss at 1 year postpartum | 1 year
  Postpartum weight loss (from last prenatal visit weight) at 1 year postpartum as a proportion of weight gained during pregnancy
Return to pre-pregnancy weight | 6 months
  Proportion of women who return to pre-pregnancy weight at 6 months postpartum
Return to pre-pregnancy weight | 1 year
  Proportion of women who return to pre-pregnancy weight at 1 year postpartum
Changes in blood pressure | 6 months
  Systolic and diastolic blood pressure at 6 months postpartum
Changes in blood pressure | 1 year
  Systolic and diastolic blood pressure at 1 year postpartum
Change in sedentary time | 6 months
  Change in self-reported sedentary time from study enrollment and study completion (completion of the study intervention). Decreased sedentary time means better outcomes.
Change in physical activity as assessed by self-reported physical activity survey | 6 months
  Change in self-reported physical activity from study enrollment and study completion as assessed by self-reported physical activity survey (Days per week exercised, length of exercise sessions). Increased physical activity means a better outcome.
Change in physical activity as assessed by modified Duke Activity Status Index | 6 months
  Change in self-reported physical activity from study enrollment and study completion as assessed by modified Duke Activity Status Index (6 question yes/no survey, score ranges from 0-31.5). A higher score means a higher functional status.
Change in stress as assessed by self-reported stress survey | 6 months
  Change in self-reported stress from study enrollment and study completion as assessed by self-reported stress survey (3 questions on scale of 0-4 [0= Never experience stress, 4= Constant stress], Max score=12). A lower score means a better outcome.
Change in stress as assessed by American Heart Association Cardiovascular Disease Go Red Questionnaire | 6 months
  Change in self-reported stress from study enrollment and study completion as assessed by American Heart Association Cardiovascular Disease Go Red Questionnaire (11 questions on scale of 0-4 [0= None of the Time, 4= All of the Time], Max score=44). A lower score means a better outcome.
Change in self efficacy for diet | 6 months
  Change in self efficacy to eat a healthy diet from study enrollment and study completion assessed by an 8-question survey rating confidence for motivating oneself to do tasks relating to eating healthy consistently for at least 6 months (Range 1 [I could not do it] to 5 [I could do it], Max score= 40). A higher score means a better outcome.
Change in self efficacy for physical activity assessed by questionnaire | 6 months
  Change in self efficacy toward achieving and maintaining a healthy level of physical activity assessed by an 8-question survey rating confidence for motivating oneself to do tasks related to physical activity consistently for at least 6 months (Range 1 [I could not do it] to 5 [I could do it], Max score= 40). A higher score means a better outcome.
Change in cardiovascular disease knowledge assessed by American Heart Association Cardiovascular Disease Go Red Questionnaire | 6 months
  Change in knowledge on the American Heart Association Cardiovascular Disease Go Red Questionnaire (modified for the postpartum population) from study enrollment and study completion (5 questions total: 4 questions on scale of 0-4 [0= Very well informed, 4= Not at all informed], Max score=16, 16-part question about the causes of heart disease [1= Yes, 2 =No], Max score = 32). A lower score means a better outcome.
Change in quality of diet assessed by Dietary Approaches to Stop Hypertension (DASH) score | 6 months
  Change in quality of diet assessed by Dietary Approaches to Stop Hypertension (DASH) score from study enrollment and study completion (DASH score range 0 [no targets met] to 9 [all targets met]). A higher score means a better outcome.

OTHER OUTCOMES:
Percent of scheduled postpartum obstetric visits attended in each treatment group | 1 year
  Percent of scheduled postpartum obstetric visits attended by patients in each treatment group
Percent of patients who attend a primary care doctor visit in each treatment group | 1 year
  Percent of patients who attend a primary care doctor visit in the 1st postpartum year in each treatment group
Percent of patients lactating in each treatment group at 6 months postpartum | 6 months
  Percent of patients lactating in each treatment group at 6 months postpartum
Percent of patients lactating in each treatment group at 1 year postpartum | 1 year
  Percent of patients lactating in each treatment group at 1 year postpartum
Percent of patients taking prescribed medications in each treatment group | 6 months
  Percent of patients who were taking prescribed medications (as assessed by refill requests documented in Epic) in each treatment group
Percent of study visits completed by patients in the intervention arm | 6 months
  Percent of study visits (out of the nutrition consultations and EP virtual visits) completed by patients in the intervention arm
Acceptability of the intervention | 6 months
  Acceptability of the intervention among study participants as assessed by exit survey (7 questions, 0= Strongly disagree, 4= Strongly agree, Max score= 28). A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Sarma, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No